CLINICAL TRIAL: NCT07287514
Title: Role of Linoleic Acid in Cardiometabolic Health Beyond Its Lipid-lowering Effects, and Its Dietary and Pathophysiological Implications
Brief Title: Metabolic Effects of Linoleic Acid-Rich Oil Compared to a Blend Oil in Adults With Insulin Resistance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Principal Investigator, Loni Berkowitz Fiebich, Assistant Professor, Pontificia Universidad Catolica de Chile
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 230330018; 11240454 (Other Grant/Funding Number: FONDECYT - ANID - Chile)
Record Dates: First submitted 2025-11-14; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Insulin Resistance; Metabolic Disease
Keywords: linoleic acid; Insulin Resistance; omega-6 fatty acid
MeSH Terms: conditions — Insulin Resistance; Metabolic Diseases

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 1:1 ratio to one of two parallel groups:
  1. an intervention group receiving a linoleic acid-rich oil, or
  2. a control group receiving a blended oil. The study follows a single-blind, parallel-group design lasting 8 weeks.
Who Masked: Participant
Masking Description: Participants are blinded; both oils are provided in identical coded bottles to maintain masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Linoleic Acid-Rich Oil (Experimental): Participants in this group will receive a daily supplement of a linoleic acid (LA)-rich oil at a dose of 0.4 mL per kilogram of body weight per day for 8 weeks.
  Interventions: Dietary Supplement: Linoleic Acid-Rich Oil
- Blend Oil (Active Comparator): Participants in this group will receive a daily supplement of a blend oil at 0.4 mL per kilogram of body weight per day for 8 weeks.
  Interventions: Dietary Supplement: Blend Oil

INTERVENTIONS:
Dietary Supplement: Linoleic Acid-Rich Oil — Participants in the experimental group will receive a daily supplement of a linoleic acid (LA)-rich oil at a dose of 0.4 mL per kilogram of body weight per day, taken orally for 8 weeks. The oil is characterized by a high content of omega-6 polyunsaturated fatty acids, primarily linoleic acid (~60%).
  To facilitate adherence and appropriate use, participants will receive a recipe booklet encouraging the use of the oil in cold or minimally cooked preparations, or as a topping over foods. They will be instructed to avoid prolonged heating and to store the oil protected from light and at room temperature.
  The supplement will be provided in identical coded bottles to maintain single-blind conditions. Participants will be asked to maintain their usual diet and lifestyle throughout the intervention.
  Arms: Linoleic Acid-Rich Oil
Dietary Supplement: Blend Oil — Participants in the control group will receive a daily supplement of a blend oil at a dose of 0.4 mL per kilogram of body weight per day, taken orally for 8 weeks. The blend was formulated to contain approximately equal proportions of saturated, monounsaturated, and polyunsaturated fatty acids, with less than half the linoleic acid content of the LA-rich oil.
  Participants will receive a recipe booklet promoting the use of the oil in cold dishes or lightly cooked preparations, or as a dressing or drizzle over meals. They will also be instructed on proper storage away from heat and direct light.
  The supplement will be supplied in identical coded bottles to ensure blinding. Participants will maintain their usual diet and lifestyle during the intervention.
  Arms: Blend Oil

SUMMARY:
Linoleic acid (LA), the predominant omega-6 polyunsaturated fatty acid in human diets, has been associated with improved lipid metabolism and insulin sensitivity compared with saturated fats. However, its role in metabolic health remains debated due to the limited number of well-controlled intervention studies.

This randomized controlled trial aims to evaluate the metabolic effects of an LA-rich oil compared with a blended oil in adults with insulin resistance. Participants will be randomly assigned to receive either a daily supplement of LA-rich oil or a control blend oil for 8 weeks, while maintaining their usual diet and lifestyle. The primary outcome is the change in insulin resistance, assessed by the Homeostatic Model Assessment of Insulin Resistance (HOMA-IR). Secondary outcomes include changes in fasting glucose, insulin, lipid profile, inflammatory and oxidative stress markers, and body composition.

The study is designed as a single-blind, parallel-group intervention conducted at the Pontifical Catholic University of Chile. The results are expected to clarify the effects of increased dietary linoleic acid intake on insulin sensitivity and metabolic risk factors, contributing to the ongoing debate about the role of omega-6 fatty acids in cardiometabolic health.

DETAILED DESCRIPTION:
Background

Non-communicable diseases (NCDs) are among the leading causes of morbidity and mortality worldwide. A healthy diet may help reduce the risk of these conditions by modulating the availability of nutrients and metabolites. However, the underlying mechanisms are not fully understood and may even lead to misconceptions.

A common example is the widespread belief that a high intake of omega-6 polyunsaturated fatty acids (PUFAs) is harmful to health. Without strong scientific support, some have advocated limiting dietary linoleic acid (LA)-the predominant PUFA in human diets-under the assumption that it competes biochemically with omega-3 fatty acids, thereby reducing their beneficial effects. Nevertheless, meta-analyses of prospective cohort studies have shown that higher LA intake or circulating levels are associated with lower total and LDL cholesterol, reduced cardiovascular disease risk, and a lower incidence of type 2 diabetes. These findings highlight the need to reassess the biological effects of LA and its potential role in metabolic regulation. To support evidence-based dietary recommendations promoting LA intake, well-controlled intervention studies are needed to better understand its cardiometabolic effects.

Hypothesis

Elevated blood levels of linoleic acid (LA), in response to increased dietary intake, confer cardiometabolic benefits beyond lipid-lowering effects, improving insulin sensitivity and reducing cardiovascular risk in individuals with cardiometabolic risk conditions.

Objectives

The primary objective is to evaluate the effect of a short-term intervention with an LA-enriched oil on insulin sensitivity and glucose homeostasis in adults with insulin resistance.

Secondary objectives include assessing the impact of the intervention on lipid profile, circulating fatty acid composition, inflammatory status, hepatic enzymes, oxidative stress markers, and estimated cardiovascular risk in Chilean adults with insulin resistance and cardiometabolic risk conditions.

Experimental Design

This study is a randomized, single-blind, controlled, parallel-group clinical trial conducted at the Clinical Research Center (CICUC) of the Pontifical Catholic University of Chile. Eligible adults with insulin resistance will be randomly assigned in a 1:1 ratio to receive either a linoleic acid-rich oil or a blend oil for 8 weeks at a dose of 0.4 mL per kilogram of body weight per day. Fasting blood samples will be collected at baseline and at 8 weeks to assess insulin resistance (HOMA-IR), lipid profile, circulating fatty acid composition, inflammatory and oxidative stress markers (AOPP, oxidized LDL), and hepatic enzymes. Anthropometric and clinical parameters will also be recorded following standardized protocols.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 20 to 60 years.
* Insulin resistance (HOMA-IR > 2.6).
* At least one cardiometabolic risk factor: abdominal obesity (waist circumference > 90 cm in men or > 80 cm in women); low HDL-cholesterol (< 40 mg/dL in men or < 50 mg/dL in women); elevated LDL-cholesterol (> 70 / 100 / 130 mg/dL, according to estimated cardiovascular risk); or elevated blood pressure (≥ 130/85 mmHg).

Exclusion Criteria:

* Diabetes diagnosis.
* Severe psychiatric illness.
* Malabsorption disorders or previous bariatric surgery.
* Pregnancy or lactation.
* Previous clinical cardiovascular disease.
* Regular use of medications that could influence study outcomes, including:

lipid-lowering agents insulin sensitizers antihypertensive drugs anticoagulants antiretroviral therapy thyroid hormones oral corticosteroids immunosuppressants polyunsaturated fatty acid (PUFA) supplements.

* Fasting serum triglycerides ≥ 500 mg/dL or LDL-cholesterol ≥ 190 mg/dL.
* Body mass index (BMI) ≥ 35 kg/m².
* Very high blood pressure.
* Any additional condition that may limit adherence to the study.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in insulin resistance (HOMA-IR) | Baseline and 8 weeks after the start of the intervention.
  Insulin resistance will be assessed using the Homeostatic Model Assessment of Insulin Resistance (HOMA-IR), calculated from fasting glucose and fasting insulin concentrations. The primary outcome is the change in HOMA-IR from baseline to week 8 between the two study groups.

SECONDARY OUTCOMES:
Glycated hemoglobin (HbA1c) | Baseline and week 8
  HbA1c (%) will be measured to assess glucose homeostasis.
Fasting glucose | Baseline and week 8
  Fasting glucose (mg/dL) will be measured to assess glucose homeostasis.
Fasting insulin | Baseline and week 8
  Fasting insulin (µU/mL) will be measured to assess glucose homeostasis.
Lipid profile | Baseline and week 8
  Plasma concentrations (mg/dL) of total cholesterol, HDL-cholesterol, LDL-cholesterol, and triglycerides will be determined using standard enzymatic assays.
Liver enzymes | Baseline and week 8
  Hepatic function will be evaluated by measuring serum concentration (U/L) of alanine aminotransferase (ALT/GPT), aspartate aminotransferase (AST/GOT), and gamma-glutamyl transferase (GGT).
Body Weight | Baseline and week 8
  Body weight will be measured using a calibrated digital scale.
Body mass index (BMI) | Baseline and week 8
  BMI will be calculated as weight (kg) divided by height squared (m²)
Waist circumference | Baseline and week 8
  Waist circumference (cm) will be measured with a non-stretchable tape at the midpoint between the iliac crest and the lowest rib
Inflammatory markers | Baseline and week 8
  Serum levels of pro-inflammatory cytokines such as tumor necrosis factor-alpha (TNF-α) and interleukin-6 (IL-6) will be measured to assess systemic inflammation.
Oxidative stress markers | Baseline and week 8
  Advanced oxidation protein products (AOPP) and oxidized LDL (oxLDL) will be measured in plasma as indicators of oxidative stress.
Change in plasma fatty acid profile | Baseline and week 8
  The plasma fatty acid composition will be determined from fasting samples by gas chromatography. Relative and absolute concentrations of major fatty acids, including linoleic acid, arachidonic acid, and docosahexaenoic acid, will be quantified to assess changes in circulating lipid composition and adherence to the assigned oil intervention.
24-hour dietary recall | Baseline and week 8
  Two non-consecutive 24-hour food recalls will be applied by trained dietitians at baseline and during the last week of the intervention to assess nutrient intake. Nutrient intake will be analyzed using ESHA's Food Processor® Nutrition Analysis software.
Diet quality (Chilean MDI) | Baseline and week 8
  Self-reported diet quality will be assessed using the Chilean Mediterranean Dietary Index (Chilean-MDI) questionnaire. The scale ranges from 0 to 14 points, where higher scores indicate greater adherence to the Mediterranean dietary pattern, reflecting better diet quality. A score of 0 represents no adherence, and 14 represents maximum adherence.
Sleep quality (PSQI) | Baseline and week 8
  Self-reported sleep quality assessed using the Pittsburgh Sleep Quality Index (PSQI) at baseline and post-intervention. The PSQI assesses subjective sleep quality across seven components, yielding a global score from 0 to 21. Higher scores indicate poorer sleep quality, with values >5 typically reflecting clinically relevant sleep disturbances.
Physical activity (GPAQ) | Baseline and week 8
  Self-reported physical activity assessed using the Global Physical Activity Questionnaire (GPAQ) at baseline and post-intervention. GPAQ provides total physical activity expressed in MET-minutes/week, typically ranging from 0 to >10,000 MET-min/week. Higher values indicate greater overall physical activity, while lower values reflect insufficient activity.

CONTACTS AND LOCATIONS:
Overall Officials: Loni Berkowitz, PhD, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- Centro de Investigaciones Clínicas UC (CICUC) - Pontificia Universidad Católica de Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared. Only aggregated results will be made available through scientific publications and presentations.

REFERENCES:
- [Background] Berkowitz L, Echeverria G, Salazar C, Faundez C, Coe CL, Ryff C, Rigotti A. Lipidomic Signature of Healthy Diet Adherence and Its Association with Cardiometabolic Risk in American Adults. Nutrients. 2024 Nov 22;16(23):3995. doi: 10.3390/nu16233995. PMID 39683389
- [Background] Berkowitz L, Razquin C, Salazar C, Biancardi F, Estruch R, Ros E, Fito M, Corella D, Coe CL, Ryff CD, Ruiz-Canela M, Salas-Salvado J, Wang D, Hu FB, Deik A, Martinez-Gonzalez MA, Rigotti A. Sphingolipid profiling as a biomarker of type 2 diabetes risk: evidence from the MIDUS and PREDIMED studies. Cardiovasc Diabetol. 2024 Dec 18;23(1):446. doi: 10.1186/s12933-024-02505-7. PMID 39695759
- [Background] Berkowitz L, Mateo C, Salazar C, Samith B, Sara D, Pinto V, Martinez X, Calzada M, von Schultzendorff A, Pedrals N, Bitran M, Echeverria G, Ruini C, Ryff C, Rigotti A. Healthy Eating as Potential Mediator of Inverse Association between Purpose in Life and Waist Circumference: Emerging Evidence from US and Chilean Cohorts. Int J Environ Res Public Health. 2023 Nov 23;20(23):7099. doi: 10.3390/ijerph20237099. PMID 38063529
- [Background] Calderon M, Plaza G, Gomez M, Samith B, Pinto V, Martinez X, Sara D, Echeverria G, Calzada M, Berkowitz L, von Schultzendorff A, Pedrals N, Bitran M, Rigotti AG. [Limitations and opportunities for the appropriation of the Mediterranean diet in Chilean adults with diagnostic elements of metabolic syndrome]. Nutr Hosp. 2024 Feb 15;41(1):86-95. doi: 10.20960/nh.04652. Spanish. PMID 38047416
- [Background] Echeverria G, Samith B, von Schultzendorf A, Pinto V, Martinez X, Sara D, Calzada M, Pacheco J, Plaza G, Scott F, Romero J, Mateo C, Julio MV, Utreras-Mendoza Y, Binder MV, Gutierrez F, Riquelme ME, Cuevas M, Willatt R, Sanchez O, Keilendt A, Butron P, Jarufe A, Huete I, Tobar J, Martin S, Alfaro V, Olivos M, Pedrals N, Bitran M, Avalos I, Ruini C, Ryff C, Perez D, Berkowitz L, Rigotti A. Mediterranean diet and psychological well-being intervention to reverse metabolic syndrome in Chile (CHILEMED trial). Contemp Clin Trials Commun. 2023 Jun 26;35:101167. doi: 10.1016/j.conctc.2023.101167. eCollection 2023 Oct. PMID 37538196